CLINICAL TRIAL: NCT04302454
Title: Androgen Deprivation Therapy for Oligo-recurrent Prostate Cancer in Addition to radioTherapy
Acronym: ADOPT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT2019-13
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Oligometastasis; Stereotactic Body Radiation Therapy; Androgen Deprivation Therapy; Biochemical recurrence; PSMA PET/CT; Metastases-directed radiotherapy; Metastases progression-free survival
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiosurgery; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized study. A total of 280 patients will participate in this study, equally divided between both study groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy without hormonal therapy (Active Comparator): Metastase-directed radiotherapy without the addition of hormonal therapy
  Interventions: Radiation: Radiotherapy
- Radiotherapy combined with hormonal therapy (Experimental): Metastase-directed radiotherapy with the addition of of short-term hormonal therapy (6 months)
  Interventions: Radiation: Radiotherapy; Drug: Leuprorelin

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy
  Other Names: MDRT; Metastase-directed radiotherapy; SBRT; Stereotactic body radiotherapy
Drug: Leuprorelin — Hormonal therapy
  Other Names: Eligard
  Arms: Radiotherapy combined with hormonal therapy

SUMMARY:
The overall aim of this project is to test the hypothesis that the addition of ADT to metastasis-directed radiotherapy (MDRT) in well-selected PCa patients with oligo-metastatic disease prolongs the metastases progression-free survival (MPFS) compared to MDRT alone.

ELIGIBILITY:
Inclusion criteria:

1. Histologically proven initial diagnosis of adenocarcinoma of the Prostate.
2. Biochemical recurrence of prostate cancer following primary local prostate treatment (radical prostatectomy, primary radiotherapy or radical prostatectomy +/- prostate bed adjuvant salvage radiotherapy) according to the EAU guidelines 2018. BCR after surgery: PSA > 0.1ng/ml. BCR after radiotherapy: PSA nadir +2 ng/ml or 3 consequent rises in PSA level (after exclusion of possible bounce effect).
3. Minimal 1 lesion and maximum 4 lesions (bone + lymph nodes) in total, without evidence of visceral metastases.

   1. Nodal relapse (N1) in the pelvis on PSMA-PET/CT with a maximum of 4 positive lymph nodes. The upper limit of the pelvis is defined as the aortic bifurcation.
   2. Nodal relapse (M1a) on PSMA-PET/CT above the aortic bifurcation with a maximum of 3 positive lymph nodes.
   3. Bone relapse on PSMA-PET/CT with a maximum of 3 lesions.
   4. Combination of a, b, c with a maximum of 4 metastases.
4. Age > 18 years.
5. Recent PSMA-PET/CT scan within 60 days prior to randomization.
6. PSA < 10 ng/ml.
7. In case of chronic use of finasteride the PSA value should be < 5 ng/ml.
8. WHO performance state 0-2.
9. Signed informed consent prior to registration/randomization.

Exclusion criteria

1. Visceral metastases.
2. PSA ≥ 10 ng/ml.
3. PSA-doubling time ≤ 3 months.
4. ADT or chemotherapy for recurrent PCa.
5. Testosterone < 1.7 nmol/l
6. Painful metastases needed pain medication (> level 1 pain medication) .
7. Invasive active cancers other than superficial non-melanoma skin cancers.
8. Inability or unwillingness to understand the information on trial-related topics, to give informed consent or to fill out QoL questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 280 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2027-10-21 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Metastases progression-free survival (MPFS) | 2.5 years after treatment
  The primary aim of this project is to test the hypothesis that the addition of ADT to MDRT in well-selected PCa patients with oligo-metastatic disease (OM) prolongs the metastases progression-free survival (MPFS) compared to MDRT alone

CONTACTS AND LOCATIONS:
Overall Officials: S. Al-Uwini, PhD, Principal Investigator — University Medical Center Groningen
Locations (13):
- Netherlands (13):
  - Radiotherapiegroep, Arnhem, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastro Clinic, Maastricht, Limburg
  - Catharina Hospital, Eindhoven, North Brabant
  - Amsterdam UMC (Location VUmc), Amsterdam, North Holland
  - Radiotherapiegroep, Deventer, Overijssel
  - Isala, Zwolle, Overijssel
  - Radiotherapy Institute Friesland, Leeuwarden, Provincie Friesland
  - Leinden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haga Hospital, The Hague, South Holland
  - UMCG, Groningen
  - Verbeeten Institute, Tilburg

REFERENCES:
- [Derived] Janssen J, Staal FHE, Brouwer CL, Langendijk JA, de Jong IJ, van Moorselaar RJA, Schuit E, Verzijlbergen JF, Smeenk RJ, Aluwini S. Androgen Deprivation therapy for Oligo-recurrent Prostate cancer in addition to radioTherapy (ADOPT): study protocol for a randomised phase III trial. BMC Cancer. 2022 May 2;22(1):482. doi: 10.1186/s12885-022-09523-2. PMID 35501744